CLINICAL TRIAL: NCT04585256
Title: The Effect of Trendelenburg Positioning on External Cephalic Version Outcome
Brief Title: Trendelenburg Positioning and External Cephalic Version Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0145-20-RMB
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Breech Presentation of Fetus With Successful Version
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trendelenburg (Active Comparator): Women positioned in the trendelenburg position during external cephalic version.
  Interventions: Other: Trendelenburg positioning
- Control (No Intervention): Women positioned on their back during external cephalic version.

INTERVENTIONS:
Other: Trendelenburg positioning — Women positioned in the trendelenburg position prior to external cephalic version
  Arms: Trendelenburg

SUMMARY:
Women at term (over 37 weeks) that are candidates for external cephalic version will be positioned in the trendelenburg position 5 minutes prior to external cephalic version performance and during the procedure. The control group will not be positioned differently than usual. We will evaluate external cephalic version success and compare the 2 groups.

DETAILED DESCRIPTION:
This is a randomized controlled trial that is designed to compare external cephalic version success between women positioned in the trendelenburg position 5 minutes prior to external cephalic version performance and during the procedure and a control group of women that will lie on their back without special positioning.

The women that are eligible for participation will receive a thorough explanation and will sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Women interested in having external cephalic version at a gestational age of 37+0/7 or more.

Exclusion Criteria:

* Age 18 and under.
* Women with a body mass index 35 or higher.
* Women with a previous cesarean section.
* Women with premature rupture of membranes.
* Women with vaginal bleeding.
* Women with a previously failed external cephalic version.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 180 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
External cephalic version success | Up to 10 minutes from the beginning of external cephalic version.
  The rate of successful external cephalic version

SECONDARY OUTCOMES:
Pain | Up to 2 hours from the beginning of external cephalic version.
  Visual analog scale scoring from 0-10 during and following the procedure.
Placental abruption | Up to 1 week from the beginning of external cephalic version.
  Rate of clinical placental abruption
Vaginal delivery | Up to 4 weeks from the beginning of external cephalic version.
  Rate of vaginal deliveries
Cesarean delivery | Up to 4 weeks from the beginning of external cephalic version.
  Rate of cesarean deliveries

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No